CLINICAL TRIAL: NCT01019187
Title: Cognitive Behavioral Therapy +/- Armodafinil for Insomnia and Fatigue Following Chemotherapy
Brief Title: Cognitive Behavioral Therapy With or Without Armodafinil in Treating Cancer Survivors With Insomnia and Fatigue After Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: UPCC 19108
Record Dates: First submitted 2009-11-13; First posted 2009-11-24 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Therapeutics; Modafinil; Medication Therapy Management; Mental Status and Dementia Tests

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Arm I (Placebo Comparator): Patients receive oral placebo twice daily for 47 days.
  Interventions: Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Placebo; Procedure: Fatigue Assessment and Management
- Arm II (Experimental): Patients receive oral armodafinil twice daily for 47 days.
  Interventions: Procedure: Sleep Disorder Therapy; Drug: Armodafinil; Procedure: Quality-of-life assessment; Other: Questionnaire Administration; Procedure: Fatigue Assessment and Management; Procedure: Management of Therapy
- Arm III (Experimental): Patients receive oral placebo twice daily for 47 days. Patients undergo cognitive behavioral therapy for insomnia comprising sleep restriction therapy, stimulus control instruction, sleep hygiene guidelines, and a session of cognitive therapy for 7 weeks.
  Interventions: Procedure: Sleep disorder therapy; Procedure: cognitive assessment; Procedure: Quality of Life assessment; Other: Questionnaire Administration; Other: Placebo; Procedure: Fatigue assessment and management; Procedure: Management of therapy and complications
- Arm IV (Experimental): Patients receive oral armodafinil twice daily for 47 days. Patients undergo cognitive behavioral therapy for insomnia as in Arm III for 7 weeks.
  Interventions: Procedure: Sleep disorder therapy; Drug: Armodafinil; Procedure: Cognitive Assessment; Procedure: Quality of Life Assessment; Other: Questionnaire Administration; Procedure: Fatifue assessment and management

INTERVENTIONS:
Procedure: Quality-of-Life Assessment — Ancillary Studies
  Arms: Arm I
Other: Questionnaire Administration — Ancillary Studies
  Arms: Arm I
Other: Placebo — Given orally
  Other Names: PLCB
  Arms: Arm I
Procedure: Fatigue Assessment and Management
  Other Names: Fatigue Assessment/Management
  Arms: Arm I
Procedure: Sleep Disorder Therapy
  Other Names: Sleep disorders therapy
  Arms: Arm II
Drug: Armodafinil — Given orally
  Other Names: Nuvigil
  Arms: Arm II
Procedure: Quality-of-life assessment — Ancillary studies
  Other Names: Quality of Life assessment
  Arms: Arm II
Other: Questionnaire Administration — Ancillary Studies
  Arms: Arm II
Procedure: Fatigue Assessment and Management
  Other Names: Fatigue Assessment and Mangement
  Arms: Arm II
Procedure: Management of Therapy
  Other Names: Complications of therapy management
  Arms: Arm II
Procedure: Sleep disorder therapy
  Arms: Arm III
Procedure: cognitive assessment
  Arms: Arm III
Procedure: Quality of Life assessment — Ancillary Studies
  Arms: Arm III
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm III
Other: Placebo — Given orally
  Other Names: PLCB
  Arms: Arm III
Procedure: Fatigue assessment and management
  Arms: Arm III
Procedure: Management of therapy and complications
  Other Names: Compllications of therapy management
  Arms: Arm III
Procedure: Sleep disorder therapy
  Other Names: sleep disorders therapy
  Arms: Arm IV
Drug: Armodafinil — Given orally
  Other Names: Nuvigil
  Arms: Arm IV
Procedure: Cognitive Assessment
  Arms: Arm IV
Procedure: Quality of Life Assessment — Quality of Life Assessment
  Other Names: Ancillary studies
  Arms: Arm IV
Other: Questionnaire Administration — Ancillary Studies
  Arms: Arm IV
Procedure: Fatifue assessment and management
  Other Names: Fatigue Assessment/management
  Arms: Arm IV

SUMMARY:
RATIONALE: Sleep disorder counseling may reduce fatigue and insomnia as well as improve the well-being and quality of life of cancer survivors. Armodafinil may help relieve insomnia and fatigue in patients with cancer after chemotherapy. PURPOSE: This randomized phase II trial is studying how well cognitive behavioral therapy with or without armodafinil works in treating cancer survivors with insomnia and fatigue after chemotherapy.

DETAILED DESCRIPTION:
Detailed DescriptionOBJECTIVES:

I. To determine if one or more of the intervention strategies (i.e., CBT-I, armodafinil, or both), when compared to a placebo only group, reduce insomnia in cancer patients following the conclusion of chemotherapy and/or radiation therapy.

II. To determine if one or more of the intervention strategies (i.e, CBT-I, armodafinil, or both), when compared to a placebo only group, reduce fatigue in cancer patients following the conclusion of chemotherapy and/or radiation therapy.

III. To determine if one or more of the intervention strategies (i.e., CBT-I, armodafinil, or both), when compared to a placebo only group, improve QOL in cancer patients following the conclusion of chemotherapy and/or radiation therapy.

OUTLINE: Patients are randomized to 1 of 4 treatment arms (cognitive behavioral therapy, armodafinil, both, or neither).

After completion of study treatment, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of cancer
* Be able to understand written and spoken English
* Be able to swallow medication
* Have preferred sleep phase between 7:30 pm and 11:00 am
* Be willing to discontinue any medications /OTCs/Herbals for sleep for the 11-week study period
* Be presumed to be in a state of cancer remission; use of tamoxifen, an aromatase inhibitor, and/or Herceptin is permitted
* Self-report problems with insomnia for at least three months and that the insomnia began or got worse with the onset of cancer or treatment
* At least one month must have passed since completion of chemotherapy and/or radiation treatment
* Report insomnia on the SDS-CL at a frequency of at least 3 days a week

Exclusion Criteria:

* Have ever taken modafinil or armodafinil had CBT-I therapy (CBT-I therapy for the sake of this protocol will be defined as any cognitive behavioral-based treatment for insomnia that includes a sleep restriction component)
* Have an unstable medical or psychiatric illness (Axis I- current or within the last 5 years)
* Have a history of seizures or severe headaches, or uncontrolled cardiac disease or hypertension
* Be presently taking an anticoagulant or a corticosteroid
* Have taken amphetamines (e.g., methylphenidate, pemoline [Cylert] or similar psycho stimulants) within the past 30 days
* Be currently pregnant or nursing
* Have a history of substance abuse, or meet criteria for current alcohol abuse or dependence as assessed by a CAGE test score >= 2 or an Alcohol Use Disorders Identification Test (AUDIT) score >= 13
* Have surgery planned within the study period
* Have ever been diagnosed with sleep apnea or have sleep apnea as indicated by endorsing either question 11 (I wake up choking or gasping for air) or question 12 (My bed partner has noticed that I seem to stop breathing) on the Sleep Disorders Symptom Check at the "Often" or "Frequently" level
* Have serious RLS/PLMs indicated by endorsing two or more items associated with RLS/PLMs on the Sleep Disorders Symptom Check at the "Frequently" level

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Severity of insomnia as assessed by the insomnia severity index and daily sleeep diaries.
Fatigue as assessed by the brief fatigue index
Adverse Events | Mid-point and end of treatment

SECONDARY OUTCOMES:
Fatigue as assessed by the functional assessment of chronic illness therapy-fatigue
Sleep latency, wake after sleep onset, and total sleep time

CONTACTS AND LOCATIONS:
Overall Officials: Michael Perlis, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811